CLINICAL TRIAL: NCT06303453
Title: Comparative Effects of Balance and Resisted Training on Pain and Balance In Patients With Diabetic Peripheral Neuropathy.
Brief Title: Comparative Effects of Balance and Resisted Training in Diabetic Peripheral Neuropathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0291
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic Peripheral Neuropathy; Balance Training; Resisted Training; Pain Management; Rehabilitation Exercises
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as assessor of the study would be kept blind of the treatment groups to which patient will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (BALANCE EXERCISES) (Experimental): Group A will receive a session of balance exercises for 45 minutes.Treatment session will be given for 3 days per week for 8 weeks.This balance exercise program consist of three phases.Warm-up phase(5 minutes,after warm-up phase 35 minutes balance exercises then cooling phase (5 minutes).
  Interventions: Other: Balance exercises
- GROUP B (RESISTED EXERCISES) (Experimental): Group B will receive a session of resisted exercises for 45 minutes.Treatment session will be given for 3 days per week for 8 weeks.This resisted exercises program consist of three phases.Warm-up phase(5 minutes,after warm-up phase 35 minutes balance exercises then cooling phase (5 minutes).
  Interventions: Other: Resisted exercises

INTERVENTIONS:
Other: Balance exercises — Balance exercises includes active movements (flexion, extension, abduction, adduction) of one upper extremity and lower extremity, trunk movements (bending forward and rotation), raising heel, raising toes and raising heel. Every move in each session will be hold for 30 seconds. The part B comprises of training i.e., holding positions in standing posture which include moving the ball up and down in a straight line with two upper extremities, moving the ball up and down in an oblique line with two upper extremities, moving the ball forward and backward with left and right lower extremities, moving the ball laterally with left and right lower extremities, throwing the ball against the wall with hand and throwing the ball against the wall with foot.
  Arms: GROUP A (BALANCE EXERCISES)
Other: Resisted exercises — The resistance training protocol include shoulder flexion and extension with 1 kg weight, shoulder pulley with 2 kg weight, arm curls with 1 kg weight, wall push-ups, bridging, hip abduction and adduction against resistance band, knee extensions and flexion in sitting position with resistance applied by contralateral limb, knee adduction and abduction with resistance band, mini squats, strengthening exercise for toes flexor and extensor (22), resisted inversion and eversion and straight leg raise (SLR) with 1 kg ankle weight (10).
  Every move in each session comprises of 2 sets of 3 reps each and 1 set will be added at 4th and 8th week.
  Arms: GROUP B (RESISTED EXERCISES)

SUMMARY:
The aim of this study is to determine comparative effects of balance and resisted training on pain and balance in patients with daibetic peripheral neuropathy.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted at Mumtaz Bakhtawar Hospital in 7 months after the approval of synopsis. The sample size for this trial will be 58 patients with DPN. Participants those meet inclusion criteria will be randomly allocated into two groups using online randomization tool, 29 participants will be assigned to Group A which will receive Balance training exercises for 35 minutes and Group B will receive Resistance Training exercises for 45 minutes. Each participant will receive intervention for 3 alternate days per week for 8 weeks.

The Michigan neuropathy screening instrument will be used for the assessment of DPN symptoms scores at baseline. Balance will be evaluated using the De Morton mobility index (DEMMI) test, while painDIRECT tool will be utilized to measure pain. The data will be entered and analyzed using SPSS version 24 for windows software.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with DNP with score ≥ 2.5 on Michigan neuropathy screening instrument of both genders.
2. Age between 40 to 65 years.
3. Patients having the minimum history of diabetes is 7 years.
4. History of mild to moderate neuropathy . The patients ability to do resistance and aerobic exercises.

Exclusion Criteria:

1. History of taking anti-inflammatory drugs.
2. History of recent surgical operations of joints in lower extremities.
3. Patients suffering from musculoskeletal disorders such as rheumatoid arthritis and myopathy.
4. Patients having any disability, fracture, or dislocation of at least six months before the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Michigan neuropathy screening instrument | 8th week
  This screening tool consists of two sections: Section A, self-administered by the patient, involves 15 yes/no questions about clinical symptoms, and Section B is based on a clinical evaluation. Positive and negative sensory symptoms, cramps, muscle weakness, foot ulcers, cracks, and amputation are assessed.
De Morton mobility index test | 8th week
  It consists of 15 items covering a broad spectrum of mobility levels and it has shown satisfactory Clinometric properties (30). In this method, the static balance is measured on one leg and two legs, as well as at the closing of the eyes; on the other hand, the dynamic balance is measured and evaluated when the patient jumps and moves four steps back.
PainDETECT Tool | 8th week
  painDETECT scale to detect diabetic neuropathic pain which includes symptom questioning and also the type, severity and the radiation of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PhD-PT, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No